CLINICAL TRIAL: NCT04005365
Title: Efficacy and Safety of Propranolol Combined With Neoadjuvant Chemotherapy in Stage III-IV Gastric Cancer: an Open-lable, Single-arm Study
Brief Title: Clinical Study of Propranolol Combined With Neoadjuvant Chemotherapy in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yijing He (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor-Investigator, Yijing He, Associate Professor, Central South University
Organization: Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/prop/GC/CSU
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer
Keywords: propranolol; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prop+neochemo (Experimental)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — add propranolol in gastric cancer patients who need to receive preoperate chemotherapy

SUMMARY:
At the cellular and animal level, we found that propranolol can inhibit the proliferation and invasion of gastric cancer cells. Further, we want to explore the efficacy and safety of propranolol in the treatment of gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent.
2. age 18 to 75;Confirmed as a primary gastric adenocarcinoma patient by imaging and histology or cytology;
3. Patients with advanced gastrointestinal cancer who have received no prior chemotherapy or radiotherapy for malignant tumors;
4. Patients with Eastern Cooperative Oncology Group Performance Status of 0 or 1.
5. Patients with a life expectancy of at least three months.;
6. Organ function and hematopoietic function must meet the following requirements: hemoglobin (HGB) ≥ 90g / L; white blood cell count (WBC) ≥ 3 × 10 ^ 9 / L; absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L Platelet count (PLT) ≥ 100 × 10 ^ 9 / L; total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase ( ALT)≤2.5×ULN; if abnormal liver function is due to tumor liver metastasis, AST or ALT≤5×ULN; serum creatinine (Cr)≤1.5×ULN; international normalized ratio (INR) or plasma prothrombin time ( PT) ≤ 1.5 × ULN.
7. Systolic blood pressure 90-140mmHg, diastolic blood pressure 60-90mmHg, heart rate 60-100bpm.
8. No previous cardiovascular and cerebrovascular diseases, and exclusion of atrioventricular block by 24-hour ambulatory electrocardiography;
9. subjects must agree to take effective contraceptive measures between the subject and the partner after signing the informed consent, during the study period and within 5 months after the last dose.

Exclusion Criteria:

1. There are clinical symptoms or diseases of the heart that are not well controlled, such as uncontrolled high blood pressure, unstable angina, or myocardial infarction within 6 months prior to enrollment, or poorly controlled arrhythmias (including QTc ( men ≥ 450ms , female ≥ 470ms, QTc interval calculated by Fridericia formula), cardiogenic shock, heart block (II-III degree atrioventricular block), severe or acute heart failure, sinus bradycardia, need continuous oxygen Treated severe respiratory diseases;
2. Subjects with symptomatic autoimmune diseases [such as, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, decreased thyroid function; The tester has vitiligo or has completely relieved asthma in childhood, and can be included without any intervention after adulthood; asthma that requires bronchodilators for medical intervention cannot be included]
3. Patients with other malignant tumors within 5 years prior to enrollment, in addition to appropriate treatment of cervical carcinoma in situ, cured skin basal cell carcinoma;
4. Immunodeficiency, such as a patient with HIV infection or other acquired, congenital immunodeficiency disease, or a history of organ transplantation
5. Patients with active tuberculosis infection by medical history or CT examination, or a history of active tuberculosis infection within 1 year prior to enrollment, or patients with a history of active tuberculosis infection more than 1 year without formal treatment;
6. Patients with tumor brain metastasis and bone marrow metastasis
7. Patients who participated in other drug clinical studies within 4 weeks;
8. Patients with history of hypersensitivity to any drugs in this study;
9. Identified as neurological or psychiatric disorders, such as epilepsy, dementia, poor compliance;
10. Alcohol abuse, drug abuse in the past year;
11. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA (HBV DNA) > 10 ^ 3 copies / mL, or hepatitis C virus antibody positive; syphilis positive;
12. Subjects had active infection or unexplained fever >38.5 degrees during Screening period before the first dose (according to the researcher, the subject can be enrolled due to fever generated by the tumor.);
13. Clinical symptoms of ascites or pleural effusion, requiring therapeutic puncture or drainage;
14. Female patients who are pregnant or lactating, or planning to become pregnant or lactating;
15. Other patients who are considered to be unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Preoperative assessment
  CR+PR

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No